CLINICAL TRIAL: NCT02281981
Title: The Effects of Repeated Bouts of Downhill Running and Curcumin Supplementation on Arterial Stiffness During Recovery
Acronym: Cur
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project abandoned
Sponsor: University of Prince Edward Island (Other)
Collaborators: OmniActive Health Technologies (Industry)
Responsible Party: Principal Investigator, Dr. Jamie Burr, Assistant Professor, University of Prince Edward Island
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Curcumin
Record Dates: First submitted 2014-10-29; First posted 2014-11-04 (Estimated); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Vascular Stiffness
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curcumin supplement (Experimental): 200 mg, curcuminoids, 7d of supplementation in capsular form
  Interventions: Dietary Supplement: Curcumin
- Placebo (Placebo Comparator): sucrose, capsular
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin — 333mg CurcuWin OAHTCUR002-2014
  Other Names: Tumeric extract
  Arms: Curcumin supplement
Dietary Supplement: Placebo — OAHTCUR005-2014
  Arms: Placebo

SUMMARY:
Arterial Stiffness: As a recognized independent indicator of cardiovascular risk, maintaining low levels of arterial stiffening is important to cardiovascular health. Increases in arterial stiffening results in elevated systolic and mean pressure and it is correlated with various cardiovascular conditions such as left ventricular hypertrophy, ischaemic heart disease, and myocardial infarction. In contrast, decreased arterial stiffness improves ventricular-vascular coupling, ejection fraction, and cardiac output. Arterial stiffness is linked to inflammation and oxidative stress. Both inflammation and oxidative stress are elevated during DOMS (delayed onset muscle soreness), a state brought on by muscle damage often incurred during strenuous exercise. Recent studies have shown that a single bout of eccentric exercise can produce acute arterial stiffness during recovery. However, anti-oxidants/anti-inflammatories may be effective in reducing the extent of damage by decreasing oxidation and inflammation. Curcumin is a powerful antioxidant that could act as an anti-inflammatory and diminish the effects of the downhill run. In addition, eccentric damage generates a prophylactic protection lasting up to six weeks. The nature of the downhill run is primarily eccentric in nature. Therefore, repeated bouts may have diminished DOMS development. Any reduction in stress by either the prophylactic repeated bout effect or the Curcumin supplement, should attenuate the increase in arterial stiffness due to the reduction in inflammation.

DETAILED DESCRIPTION:
Baseline Participants will report to the lab on day one to have basic anthropometry and clinical measures performed. Following measures of height, weight, blood pressure, blood lipids (fasting glucose), creatine kinase, high sensitivity C-reactive protein (HS-CRP) and interleukin-6 (IL-6) participants will be allowed to eat a small standardized snack. Participants will then have measures of baseline muscle soreness and leg strength measured prior to a VO2max test on a cycle ergometer.

Muscle Soreness will be measured using a standard 10cm analogue scale and girth of the thigh will be recorded to account for possible alterations owing to local inflammation/oedema./ Creatine Kinase (CK) will be tracked as a measure of damage.

The test termination criteria for the VO2max will include: volitional fatigue, a participant rating of perceived exertion of 19-20 (on a scale from 0-20), a plateau in O2 uptake with increasing workload, or and RER of >1.15. The VT of each participant will be noted to compare with values post- training.

Testing Day 2 - This day will occur at least 1 full day (48h) following VO2max testing.

Participants will arrive at the lab having consumed a standardized breakfast. Prior to the downhill run, measures of pulse wave velocity (PWV), heart rate variability (HRV), flow mediated dilatation (FMD) will be collected according to the protocols to follow. Participants will then perform a 40 minute downhill run at a grade of -12 percent using a speed that elicits a VO2 of approximately 60% of the maximum value achieved during the max test.

Arterial stiffness will be determined using a Sphygmocor CPVH pulse wave applanation tonomoter (Atcor Medical). This device measures arterial pulse waves non-invasively through the skin. By matching pulse wave arrival with heart beats (through a standard ECG tracing) and measuring the distance between points we can calculate travel time (or velocity). We will also use this same device to analyze the shape of the pulse wave, which will give us information about reflected pulse waves (and thus the stiffness of the arterial tree).

Follow-up: At 24h, 48h, and 72h post exercise, participants will return to the lab to have all of the non-exercise measures repeated (see figure 1). This will allow temporal tracking over time.

Hypotheses:

1) The anti-inflammatory potential of Curcumin supplementation should improve post-exercise recovery. 2) Repeated bouts of eccentrically biased downhill running should produce a prophylactic effect and reduce arterial stiffness and recovery time

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be male or female
* 18yr - 45yr
* Free from any known or suspected chronic conditions.
* General health and suitability to participate in an exercise/health research study will be confirmed through use of the PAR-Q+ screening questionnaire

Exclusion Criteria:

* Any participant who has a positive answer to a screening question will be required to seek physician approval prior to any physical exercise.
* Baseline arrhythmia (tachycardia (>100pbm) and systolic or diastolic hypertension (>140/90 mmHg) will also be reason for exclusion.
* During baseline anthropometric assessment we will confirm that participants all fall within a typical BMI range (20-30 kg/m2) of either "normal" weight or "overweight", but not "underweight" or "obese".
* Persons who take cardiovascular medications, metabolic medications, smoke cigarettes, excessively consume alcohol, are prone to heartburn, or have a previous diagnosis of hyperlipidemia or hyperinsulemia will also be excluded

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Arterial Stiffness | Every 24 hr up to 72hr post baseline
  This will be measured using arterial tonometry
Blood measures of inflammation and muscle damage | Every 24 hr up to 72hr post baseline
  Interleukin-6, highsensitivity C-reactive protein, Creatine Kinase

SECONDARY OUTCOMES:
Delayed onset muscle soreness | Every 24 hr up to 72hr post baseline
  Subjective analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Jamie F Burr, PhD, Principal Investigator — UPEI